CLINICAL TRIAL: NCT01699763
Title: Evaluation of Blood Glucose Meter Systems - Contour® NEXT LINK Study
Brief Title: Evaluation of Blood Glucose Monitoring Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTD-2012-007-01
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Results first posted 2013-11-28 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects with and without Diabetes (Experimental): All testing and lancing were performed by the study staff; Subjects with and without Diabetes did not perform any lancing or self-testing in this study. Study Staff lanced the fingers of subjects and tested the blood samples using three Blood Glucose Monitoring Systems (BGMS): Contour® NEXT LINK BGMS; OneTouch® UltraLink® BGMS; Nova Max Link® BGMS.
  Interventions: Device: Contour® NEXT LINK BGMS; Device: OneTouch® UltraLink® BGMS; Device: Nova Max Link® BGMS

INTERVENTIONS:
Device: Contour® NEXT LINK BGMS — Study staff performed Blood Glucose (BG) tests with capillary fingerstick blood collected from subjects with and without diabetes (up to 10% of subjects without diabetes were included). Performance of Contour® NEXT LINK BGMS was evaluated across the glucose range of the BGMSs. All meter BG results were compared with capillary plasma results obtained with a reference laboratory glucose method (YSI Glucose Analyzer).
Device: OneTouch® UltraLink® BGMS — Study staff performed Blood Glucose (BG) tests with capillary fingerstick blood collected from subjects with and without diabetes (up to 10% of subjects without diabetes were included). Performance of OneTouch® UltraLink® BGMS was evaluated across the glucose range of the BGMSs. All meter BG results were compared with capillary plasma results obtained with a reference laboratory glucose method (YSI Glucose Analyzer).
Device: Nova Max Link® BGMS — Study staff performed Blood Glucose (BG) tests with capillary fingerstick blood collected from subjects with and without diabetes (up to 10% of subjects without diabetes were included). Performance of Nova Max Link® BGMS was evaluated across the glucose range of the BGMSs. All meter BG results were compared with capillary plasma results obtained with a reference laboratory glucose method (YSI Glucose Analyzer).

SUMMARY:
The purpose of this study was to evaluate the performance of a Bayer Blood Glucose Monitoring System (BGMS) and two additional Blood Glucose Monitoring Systems (BGMS) from other companies. All meter BG results were compared with plasma results obtained with a reference laboratory glucose method (YSI Glucose Analyzer).

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the performance of a Bayer Blood Glucose Monitoring System (BGMS) and two additional Blood Glucose Monitoring Systems (BGMS) from other companies. All meter BG results were compared with plasma results obtained with a reference laboratory glucose method (YSI Glucose Analyzer). Performance of the three systems was evaluated across the glucose range of the BGMSs using capillary blood. All testing and lancing was performed by study staff and some samples were tested from subject fingertips. Additionally, some blood samples were glycolyzed to lower the glucose concentration levels and glucose solution was added to other samples to raise glucose concentration levels.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years of age or older
* Willing to complete all study procedures

Exclusion Criteria:

* Blood Borne infections like hepatitis or HIV or infections such as tuberculosis
* Hemophilia or any other bleeding disorder
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2012-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Simmons, MD, Principal Investigator — Ascensia Diabetes Care
Locations (1):
- Bayer HealthCare LLC, Diabetes Care, Mishawaka, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects With and Without Diabetes: All testing and lancing were performed by the study staff; subjects with and without diabetes did not perform any lancing or self-testing in this study. Study Staff tested the blood samples using three Blood Glucose Monitoring Systems (BGMS): Contour® NEXT LINK BGMS; OneTouch® UltraLink® BGMS; Nova Max Link® BGMS.
Period: Overall Study
Arm/Group | Subjects With and Without Diabetes
Started | 112
Completed | 112
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Subjects With and Without Diabetes
Number analyzed (Participants) | 112
Age, Continuous [Median (Full Range); unit: years] | 59 [19 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 45
Region of Enrollment [Number; unit: participants]
  United States | 112

OUTCOME MEASURES:

1. Primary Outcome: MARD (Mean Absolute Relative Difference Between BGMS Results and Reference Method Results) Across the Overall Tested Glucose Range
Description: Using the overall Blood Glucose (BG) range (34 to 561 mg/dL according to YSI subject plasma results), the Mean Absolute Relative Differences (MARD) between the BGM System readings and the YSI plasma results (BG reference) were compared. MARD is calculated from the sum of all |(BG meter)-(BG reference)|/(BG reference) assessments, divided by the number of assessments, then multiplied by 100(%). Each evaluable sample was tested on all 3 BGMS, thus the same number of BG test results was analyzed for each BGMS intervention. Lower MARD value indicates smaller difference between meter value and the reference value. Higher MARD value indicates larger difference between meter value and the reference value.
Time Frame: 8 hours
Population: Same number 333 (336-3) BG results possible for each BGMS. Staff collected 3 capillary samples from each subject - total 336 samples. Three samples from one subject were not analyzed. Subject hematocrit (58.5) was above the study evaluable limit of 55.
Measure: Mean (Standard Error); unit: Percent Difference
Units Other Than Participants: BG test results
Arm/Group | Subjects With and Without Diabetes
Number analyzed (Participants) | 111
Number analyzed (BG test results) | 333
Percent Difference
  Contour® NEXT LINK BGMS | 2.7 (0.33)
  OneTouch® UltraLink® BGMS | 10.8 (0.33)
  Nova Max Link® BGMS | 6.4 (0.33)

2. Secondary Outcome: MARD (Mean Absolute Relative Difference Between BGMS Results and Reference Method Results) in the Low Glucose Range (<=80 mg/dL)
Description: Using fresh and glycolyzed samples with YSI plasma Blood Glucose (BG) ≤80 mg/dL, the Mean Absolute Relative Differences (MARD) between the BGM System readings and the YSI subject plasma results (BG reference) were compared. MARD is calculated from the sum of all |(BG meter)-(BG reference)|/(BG reference) assessments, divided by the number of assessments, then multiplied by 100(%). Each evaluable sample was tested on all 3 BGMS, thus the same number of BG test results was analyzed for each BGMS intervention. Lower MARD value indicates smaller difference between meter value and the reference value. Higher MARD value indicates larger difference between meter value and the reference value.
Time Frame: 8 hours
Population: Same number (107) of BG results was possible for each BGMS. Staff collected 3 capillary samples from each subject (total 333), of which 107 samples were less than or equal to 80 mg/dL.
Measure: Mean (Standard Error); unit: Percent Difference
Units Other Than Participants: BG test results
Arm/Group | Subjects With and Without Diabetes
Number analyzed (Participants) | 111
Number analyzed (BG test results) | 107
Percent Difference
  Contour® NEXT LINK BGMS | 2.63 (0.69)
  OneTouch® UltraLink® BGMS | 14.92 (0.69)
  Nova Max Link® BGMS | 8.81 (0.69)

3. Secondary Outcome: MARD (Mean Absolute Relative Difference Between BGMS Results and Reference Method Results) in the High Glucose Range (>180 mg/dL)
Description: Using samples with YSI plasma Blood Glucose (BG) >180 mg/dL, the Mean Absolute Relative Differences (MARD) between the BGM System readings and the YSI subject plasma results (BG reference) were compared. MARD is calculated from the sum of all |(BG meter)-(BG reference)|/(BG reference) assessments, divided by the number of assessments, then multiplied by 100(%). Each evaluable sample was tested on all 3 BGMS, thus the same number of BG test results was analyzed for each BGMS intervention. Lower MARD value indicates smaller difference between meter value and the reference value. Higher MARD value indicates larger difference between meter value and the reference value.
Time Frame: 8 hours
Population: Same number (106) of BG results was possible for each BGMS. Staff collected 3 capillary samples from each subject (total 333), of which 106 samples were greater than 180 mg/dL.
Measure: Mean (Standard Error); unit: Percent Difference
Units Other Than Participants: BG test results
Arm/Group | Subjects With and Without Diabetes
Number analyzed (Participants) | 111
Number analyzed (BG test results) | 106
Percent Difference
  Contour® NEXT LINK BGMS | 2.66 (0.76)
  OneTouch® UltraLink® BGMS | 8.76 (0.76)
  Nova Max Link® BGMS | 4.52 (0.76)

ADVERSE EVENTS:
Arm/Group | Subjects With and Without Diabetes
Serious Adverse Events (participants affected / at risk) | 0/112
Other Adverse Events (participants affected / at risk) | 2/112
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With and Without Diabetes (N=112)
hypoglycemia (Endocrine disorders) | 2 (2) — Adverse event was mild, anticipated, non-device related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes